CLINICAL TRIAL: NCT03522675
Title: Skin Prick Test in Healthy Volunteers of Any Sex, to Investigate the Potential Allergy to NeoMatriXTM Wound Matrix
Brief Title: NeoMatriX Wound Matrix Collagen Dressing Skin Prick Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeXtGen Biologics, Inc. (Industry)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL-18002
Record Dates: First submitted 2018-04-19; First posted 2018-05-11 (Actual); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Allergy Skin; Allergy; Dermatitis, Allergic Contact
MeSH Terms: conditions — Hypersensitivity; Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- NeoMatriX and Two Comparators (Other): NeoMatriX Wound Matrix Collagen Dressing 8mm disc Histamine positive control (0.1mL) Normal saline negative control (0.1mL)
  Interventions: Device: NeoMatriX Wound MatriX Collagen Dressing

INTERVENTIONS:
Device: NeoMatriX Wound MatriX Collagen Dressing — Collagen wound dressing

SUMMARY:
The objective of this study is to investigate the potential of NeoMatriXTM Wound Matrix to cause an allergic response to healthy volunteers using a skin prick test.

DETAILED DESCRIPTION:
Using a minimally invasive skin prick test, the test material, positive control, and negative control are applied to the forearm using a prick test. The test area is observed after 15 minutes, 6 hours, and again at 1-2 days after the initial prick test. The skin will be examined for a reaction such as a wheal and/or a flare, a flare alone is not clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged at least 18 years.
* Completed written informed consent and receive a copy of their executed ICF.
* Volunteers must be capable of understanding and following directions in English.

Exclusion Criteria:

* Pregnancy or lactation;
* Inadequate or non-existent contraception (women of child bearing potential only);
* A current skin disease;
* Heavy alcohol consumption;
* Current use or history of repeated use of recreational drugs;
* Recent illness prior to test;
* Significant past medical history of diseases to potentially effect study results;
* Current treatment of allergy;
* A history of multiple drug hypersensitivity;
* Concurrent medication likely to affect the response to the test articles or confuse the results of the study;
* Known sensitivity to the test articles;
* Participation in a repeat insult patch test (RIPT), skin prick test (SPT) or follow-up work within the last month;
* Sensitization or questionable sensitization in a skin test;
* Recent immunization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo Clinical and Translational Research Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NeoMatriX and Two Comparators
Started | 22
Completed | 20
Not Completed | 2
Not completed — Screen fail | 1
Not completed — Non-reactive to histamine | 1

BASELINE CHARACTERISTICS:
Arm/Group | NeoMatriX and Two Comparators
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.35 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Wheal Formation
Description: Wheal formation is defined as a raised, pale, itchy formation (allergic reaction) on the skin's surface. A positive (+) allergic response would be indicated by the NeoMatriXTM Wound Matrix producing a wheal >3 mm of the positive control (histamine).
Time Frame: 15 minutes
Measure: Mean (Full Range); unit: mm
Groups:
- NeoMatriX Alone: NeoMatriX Wound Matrix Collagen Dressing 8mm disc
  NeoMatriX Wound MatriX Collagen Dressing: Collagen wound dressing
- Positive Control: Histamine positive control (0.1mL)
- Negative Control: Normal saline negative control (0.1mL)
Arm/Group | NeoMatriX Alone | Positive Control | Negative Control
Number analyzed (Participants) | 20 | 20 | 20
mm | .85 [0 to 3.5] | 6.68 [4.5 to 11] | .2 [0 to 3]

2. Other Pre Specified Outcome: Wheal Formation
Description: as for outcome 1
Time Frame: 6 hrs
Measure: Mean (Full Range); unit: mm
Arm/Group | NeoMatriX Alone | Positive Control | Negative Control
Number analyzed (Participants) | 20 | 20 | 20
mm | 0 [0 to 0] | 0.1 [0 to 1] | 0 [0 to 0]

3. Other Pre Specified Outcome: Wheal Formation
Description: as for outcome 1
Time Frame: 2 days
Measure: Mean (Full Range); unit: mm
Arm/Group | NeoMatriX Alone | Positive Control | Negative Control
Number analyzed (Participants) | 20 | 20 | 20
mm | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- Histamine + NeoMatriX: NeoMatriX Wound Matrix Collagen Dressing 8mm disc Histamine positive control (0.1mL)
- Saline + NeoMatriX: NeoMatriX Wound Matrix Collagen Dressing 8mm disc
  Normal saline negative control (0.1mL)
Arm/Group | NeoMatriX Alone | Histamine + NeoMatriX | Saline + NeoMatriX
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03522675/Prot_000.pdf